CLINICAL TRIAL: NCT04770467
Title: A Phase 2, Randomized, Single-blinded, Placebo-controlled Study to Evaluate the Safety and Efficacy of Human Monoclonal Antibodies, BRII-196 and BRII-198, Administered by Intravenous Infusion for the Treatment of COVID-19 Patients
Brief Title: A Safety and Efficacy Study of Human Monoclonal Antibodies, BRII-196 and BRII-198 for the Treatment of Patients With COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study will no longer move forward due to recent changes in COVID-19 cases in Hong Kong.
Sponsor: Brii Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Organization: Brii Biosciences Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRII-196-198-002
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: COVID-19 phase 2; monoclonal antibody
MeSH Terms: conditions — COVID-19 | interventions — amubarvimab; romlusevimab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BRII-196 and BRII-198 in adult subjects with severe COVID-19 (Experimental)
  Interventions: Drug: BRII-196 and BRII-198
- Placebo in adult subjects with severe COVID-19 (Placebo Comparator)
  Interventions: Drug: Placebo
- BRII-196 and BRII-198 in adult subjects with mild-moderate COVID-19 (Experimental)
  Interventions: Drug: BRII-196 and BRII-198
- Placebo in adult subjects with mild-moderate COVID-19 (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BRII-196 and BRII-198 — BRII-196 and BRII-198 given by intravenous administration
  Arms: BRII-196 and BRII-198 in adult subjects with mild-moderate COVID-19; BRII-196 and BRII-198 in adult subjects with severe COVID-19
Drug: Placebo — Placebo given by intravenous administration
  Arms: Placebo in adult subjects with mild-moderate COVID-19; Placebo in adult subjects with severe COVID-19

SUMMARY:
This study is to evaluate the safety, efficacy and pharmacokinetics profile of human monoclonal antibodies, BRII-196 and BRII-198 compared with placebo in patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Subject ≥ 18 years, signing the informed consent.
* SARS-CoV-2 infection by PCR ≤ 7 days
* One or more of COVID-19 related symptoms or measured fever present within 48 hours prior to study entry (subjects with mild-moderate COVID-19)

Exclusion Criteria:

* Recurring COVID-19 patients.
* Subjects with any unstable conditions, a history of significant hypersensitivity, or known allergy to components of the investigational agent
* Receipt of convalescent COVID-19 plasma, SARS-CoV-2 mAb treatment, SARS-CoV-2 vaccine, or other investigational treatments prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Day 29
Incidence of serious adverse events (SAEs) | up to Day 29
Change from pre-dose baseline in RBC count | Day 29
Change from pre-dose baseline in WBC count | Day 29
Change from pre-dose baseline in Platelets count | Day 29
Change from pre-dose baseline in Hemoglobin result | Day 29
Change from pre-dose baseline in Creatine kinase result | Day 29
Change from pre-dose baseline in Alanine aminotransferase (ALT) result | Day 29
Time-weighted average changes in SARSCoV-2 RNA levels in nasopharyngeal swabs from baseline to Day 8 | Day 8

SECONDARY OUTCOMES:
Duration of COVID-19 related symptoms through Day 29 among subjects with mild-moderate COVID-19 | up to Day 29
Proportion of subjects who have mild-moderate COVID-19 and develop severe COVID-19 after randomization | up to 72 weeks
Assessment of PK parameters: maximum serum concentration observed (Cmax) | up to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Yao Zhang, MD, Study Director — Brii Biosciences, Inc.
Locations (1):
- Investigative Site 1, Hong Kong, China

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343